CLINICAL TRIAL: NCT06534073
Title: Identification of Baropodometric Patterns Associated with Metatarsalgia and Custom Design of Its Three-dimensional Element of Discharge to Integrate It in Stockings or Socks
Brief Title: Baropodometric Patterns Associated with Metatarsalgia
Acronym: IMEDESCAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Pedro V. Munuera-Martínez, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N2009020
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-01

CONDITIONS: Metatarsalgia
MeSH Terms: conditions — Metatarsalgia | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Socks (Experimental): The intervention will be the daily use of socks with the integration of the customized orthotic element.
  Interventions: Device: Socks
- Standard device (Other): The intervention will be the daily use of external orthotic elements (to be put on and taken off daily) and of standard manufacture.
  Interventions: Device: Standard device
- Foot orthoses (Other): The participants will receive completely personalized plantar supports integrating the relief element.
  Interventions: Device: Foot orthoses

INTERVENTIONS:
Device: Socks — Plantar orthotic elements will be designed, according to the participants' previous baropodometric pattern, to alleviate pathological plantar pressure. These elements will be integrated into commonly worn items by patients, such as stockings or socks.
  Arms: Socks
Device: Standard device — Removable device of digital alignment to stabilize and unload the affected metatarsophalangeal joint. They do not require frequent replacement as they are washable and reusable elements.
  Arms: Standard device
Device: Foot orthoses — Custom-made foot orthoses.
  Arms: Foot orthoses

SUMMARY:
The therapeutic plan for certain pathologies in the adult population typically includes the performance of moderate physical activity aimed at preventing cardiovascular risk due to sedentary lifestyle, improving muscle tone and balance to prevent falls, enhancing bone health, and maintaining proper functional and mental health state. However, this activity can be hindered by pain arising from musculoskeletal injuries of low or moderate significance. One such injury is metatarsalgia, characterized by acute or chronic pain in the plantar area of the forefoot due to an overload of plantar pressure. It affects one or several central metatarsals and their respective metatarsophalangeal joints. Metatarsalgia is a highly prevalent pathology (up to 83%) in patients aged 60 or older and negatively impacts their quality of life. To alleviate plantar pressure in the affected area, metatarsal offloading devices are commonly used, which can now be integrated into socks or stockings. This integration aids in pain reduction through an everyday, easy-to-use item. However, only preliminary results of their effectiveness exist, and are in a standard model without customization for the patient's foot. Therefore, the goal is to identify different plantar pressure patterns in a sample of female patients over 55 years with metatarsalgia and design personalized three-dimensional plantar elements that can be integrated into the sock's structure to reduce over pressure and improve the clinical picture. A prior evaluation of pain (Foot Pain and Disability Index), impact on quality of life (SF-12 questionnaire), assessment of physical activity (IPAQ), and baropodometric evaluation with instrumented Pedar® insoles (Novel, Germany) will be conducted. This will characterize the patterns of plantar pain. Using 3D scanning of the foot, a personalized three-dimensional element for each plantar pain pattern will be designed to relieve this excess load, and will be integrated into the body of the sock through weaving, thermofusion, or thermosealing. This sample of patients with metatarsalgia will be randomly divided into three groups, who for a period of six months will wear the offloading sock model, personalized plantar supports with selective offloading, or a stabilizing element for the affected metatarsal head that the patient can apply and remove themselves. After these six months, plantar pain, quality of life, and physical activity levels will be re-evaluated in the three groups to determine the potential efficacy of the experimental sock compared to the best possible treatment, insoles, and another common element such as alignment devices. The offloading sock would provide a personalized solution for each patient, requiring no adaptation or frequent replacement, thus creating better adherence to treatment. The number of effective treatment usage hours would increase since socks are part of the patients' regular attire. Additionally, associated costs would be reduced, as there would be no need for frequent replacement of removable pads, stabilizing devices, or regular revisions to adjust orthopedic insoles.

ELIGIBILITY:
Inclusion Criteria:

* Female sex;
* Age ≥ 55 years;
* Experiencing moderate to severe pain in the plantar area of the forefoot;
* Presenting hyperkeratosis under the central metatarsal heads;
* Presenting pre-dislocation syndrome of the second or third metatarsophalangeal joint.

Exclusion Criteria:

* Present cognitive deterioration that impedes the proper development of the study;
* Have undergone previous osteoarticular surgeries on the feet;
* Diagnosis of rheumatoid arthritis with involvement in the metatarsophalangeal joints of the foot;
* Present symptoms compatible with Morton's neuritis;
* Use of walking aids;
* Are under treatment with insoles;
* Refuse the use of designated socks or plantar supports during the follow-up period.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Score 11 | 4 weeks
  Pain under the metatarsal heads of the feet, using the Numeric Pain Rating Score 11 (NPRS-11), in which the minimum value is 0 (no pain) and the maximum value is 10 (the worst imaginable pain).

IPD SHARING:
Plan to Share IPD: Yes
It is planned that the datasets generated during the project will be deposited in the institutional repository of the University of Extremadura and the University of Seville, whose metadata are aggregated to RECOLECTA of the Fundación Española para la Ciencia y la Tecnología (FECYT) and OpenAIRE Explore. The repository uses the generic Dublin Core metadata standard for dataset description and provides a handle as a permanent identifier. Data that contains potentially identifiable information about human subjects will not be publicly shared. And they cannot be disclosed until the patents related to this research are managed. In all activities carried out during this project, the fundamental principles of research integrity will be respected, following the Code of Good Research Practices of the University of Extremadura and the University of Seville, and all necessary procedures will be followed to comply with current data protection legislation.
Supporting Information: SAP, CSR